CLINICAL TRIAL: NCT03225170
Title: Is it Feasible?: Self-Affirmation for Hereditary Breast and Ovarian Cancer Genetic Counseling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 999917132; 17-HG-N132
Record Dates: First submitted 2017-07-20; First posted 2017-07-21 (Actual); Results first posted 2022-01-11 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2020-06-29

CONDITIONS: Breast Cancer
Keywords: Decision-Making; BRCA1; BRCA2; Genetic Counseling; HBOC
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-affirmation (SA) group (Experimental): Immediately prior to the scheduled cancer genetic counseling appointment, clients:
  1. completed standardized questionnaires on self-affirmation (SA) intervention that focused on positive values of personal importance. The SA intervention required clients to rank 11 items (artistic skills, athletics, business/money, creativity, independence, music, politics, relationships with friends and family, religious values, sense of humor, spontaneity) from most important to least important and to elaborate on one that was most important to them and why;
  2. 6-item standardized measure of anxiety questionnaire;
  3. after the genetic counseling session, clients were required to fill out a post session questionnaire
  Interventions: Behavioral: Self Affirmation (SA)
- Control group (Sham Comparator): Immediately prior to the scheduled cancer genetic counseling appointment, clients:
  1. completed similar standardized questionnaire as the SA group, with a non-affirming exercise. The non-intervention required clients to rank 11 items (artistic skills, athletics, business/money, creativity, independence, music, politics, relationships with friends and family, religious values, sense of humor, spontaneity) from most important to least important and to elaborate on the 9th ranked item and why it might be important to someone else;
  2. 6-item standardized measure of anxiety questionnaire;
  3. after the genetic counseling session, clients were required to fill out a post session questionnaire
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Self Affirmation (SA) — Clients will be asked to rank artistic skills, athletics, business/money, creativity, independence, music, politics, relationships with friends and family, religious values, sense of humor, spontaneity from most important to least important. They will then be asked to write about the item that is most important to them and why it may be important to them.
  Arms: Self-affirmation (SA) group
Behavioral: Control — Clients will be asked to rank artistic skills, athletics, business/money, creativity, independence, music, politics, relationships with friends and family, religious values, sense of humor, spontaneity from most important to least important. The control group will rank the list and be asked to write about the 9th ranked item and why it might be important to someone else.
  Arms: Control group

SUMMARY:
Background:

Some women have a high chance of developing breast and ovarian cancer because of a change in a gene that is passed within a family from one generation to the next. These women with hereditary breast and ovarian cancer (HBOC) have to make hard choices about tests and treatments. Researchers want to study how to help women to feel ready to make those choices. A kind of writing exercise might help if it is done before genetic counseling. This writing exercise is called a self-affirmation (SA) exercise. It may lead to better communication during counseling and better behavioral outcomes.

Objective:

To see if an SA exercise done before HBOC genetic counseling could improve client communication and behavior.

Eligibility:

* Clients: Adult female >=18 years of age with initial appointment for HBOC risk with genetic counselor at St. Luke's Health System
* Genetic Counselors: Genetic counselors >=18 years of age providing genetic counseling to clients at risk for HBOC

Design:

Clients will be screened by phone prior to their genetic counseling appointment.

They will arrive 15 minutes early to their appointment.

They will do a 10 to 15 minute survey and writing exercise. This includes questions about:

* Things that are important to them
* How they are feeling prior to the appointment

After their genetic counseling appointment, they will take a 10- to 15-minute follow-up survey. It can be in the office or online. It will include questions about:

* How they felt about the writing exercise
* How they felt about their genetic counseling
* If they had cancer
* If they were offered and had genetic testing

Genetic counselor participants will take a 2 to 5 minute survey after each session with a client in the study. This will include questions about how the client was in the session. They also will take a 10 to 15 minute survey at the end of the study. It will be about their opinions on the process of having their clients complete the writing exercise.

DETAILED DESCRIPTION:
The proposed study is a feasibility study to assess the viability of implementing a Self-Affirmation (SA) intervention in a Hereditary Breast and Ovarian Cancer (HBOC) genetic counseling clinic to improve client communication and behavioral outcomes. Participants will be clients and genetic counselors at the St. Luke's Hospital System HBOC clinic. This study seeks to identify outcomes that would be most informative in a large-scale research protocol. As outcomes, we will assess clients' decision self-efficacy, intention to talk with family, genetic test uptake, empowerment, and HBOC knowledge. We will also assess genetic counselors' and clients' perceived benefits, perceived harms, and acceptance of the affirmation intervention.

In this study clients will be invited to participate in an intervention before their genetic counseling appointment. The SA intervention is a short written exercise to reinforce clients' self-integrity (a global sense of personal adequacy) leading to more openness to threatening information within the genetic counseling session. Clients and genetic counselors will be surveyed to assess outcome measures and feasibility of the intervention.

Social science research has shown that when people are faced with threatening information they often seek to protect themselves and reject the threatening message. Message rejection can include minimizing the importance or discrediting the truth of the message. SA interventions aim to bolster self-integrity or esteem by focusing on aspects of participants' lives they value and thereby improving participants' self-perception and tolerance towards threatening messages. SA manipulations have been shown to increase patient communication within appointments and both intentions and actions toward behavior change.

Often in cancer genetic counseling appointments clients are confronted with the threat of having a significantly increased risk for cancers while being asked to make a decision about genetic testing. A self-affirmation intervention may facilitate greater client decision self-efficacy, empowerment, and positive behavior outcomes, such as communication with family regarding genetic risk and screening behaviors.

ELIGIBILITY:
INCLUSION CRITERIA:

Client Participants:

* Must be female, at least 18 years old
* Have an initial appointment for genetic counseling for HBOC risk at St. Luke's Health System
* Must be able to read and write in English to participate
* Pregnant women will be included

Genetic Counselor (GC) Participants:

-Must be certified GCs who see clients with an indication for HBOC related genetic counseling at St. Luke's Health System

EXCLUSION CRITERIA:

* Non-English speakers and illiterate subjects will be excluded
* Clients who are unable to provide consent will be excluded

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2020-06-29 (Actual); Study Completion 2020-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori Erby, Ph.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- St. Luke's Health System, Kansas City, Missouri, United States

REFERENCES:
- [Result] Scherr CL, Christie J, Vadaparampil ST. Breast Cancer Survivors' Knowledge of Hereditary Breast and Ovarian Cancer following Genetic Counseling: An Exploration of General and Survivor-Specific Knowledge Items. Public Health Genomics. 2016;19(1):1-10. doi: 10.1159/000439162. Epub 2015 Sep 22. PMID 26389838
- [Result] Kaphingst KA, Facio FM, Cheng MR, Brooks S, Eidem H, Linn A, Biesecker BB, Biesecker LG. Effects of informed consent for individual genome sequencing on relevant knowledge. Clin Genet. 2012 Nov;82(5):408-15. doi: 10.1111/j.1399-0004.2012.01909.x. Epub 2012 Aug 7. PMID 22694298
- [Result] Harris PR, Napper L. Self-affirmation and the biased processing of threatening health-risk information. Pers Soc Psychol Bull. 2005 Sep;31(9):1250-63. doi: 10.1177/0146167205274694. PMID 16055644
- [Result] Ferrer RA, Klein WM, Graff KA. Self-affirmation increases defensiveness toward health risk information among those experiencing negative emotions: Results from two national samples. Health Psychol. 2017 Apr;36(4):380-391. doi: 10.1037/hea0000460. Epub 2017 Feb 16. PMID 28206787

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 64 participants consented to the study, 17 participants withdrew prior to randomization and 47 participants started the study.
Groups:
- Genetic Counselor (GC): 1. Genetic Counselors (GC) provided their Standard of Care treatment, blinded to clients' enrollment in SA intervention or Control group and assessed each client's empowerment at the end of each session.
  2. GC also completed a survey at the end of the study to assess the writing exercise and the feasibility of SA for larger studies.
Period: Overall Study
Arm/Group | Self-affirmation (SA) Group | Control Group | Genetic Counselor (GC)
Started | 23 | 22 | 2
Completed | 19 | 17 | 2
Not Completed | 4 | 5 | 0
Not completed — Lost to Follow-up | 4 | 4 | 0
Not completed — Did not complete intervention/control writing exercise | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Self-affirmation (SA) Group | Control Group | Genetic Counselor (GC) | Total
Number analyzed (Participants) | 23 | 22 | 2 | 47
Age, Customized [Count of Participants; unit: Participants]
  >=18 to <65 years | 15 | 8 | 0 | 23
  >=65 years | 2 | 3 | 0 | 5
  Age Unknown (years) | 6 | 11 | 2 | 19
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 0 | 0 | 0 | 0
  Female | 23 | 22 | 0 | 45
  Gender unknown | 0 | 0 | 2 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 18 | 17 | 0 | 35
  Unknown or Not Reported | 5 | 5 | 2 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 0 | 2
  White | 16 | 17 | 0 | 33
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 5 | 2 | 11
Region of Enrollment [Number; unit: participants]
  United States | 23 | 22 | 2 | 47

OUTCOME MEASURES:

1. Primary Outcome: Test Uptake: Number of Clients Who Indicated Intention to Have Genetic Testing
Description: Intention to have genetic testing was measured with a single survey item, "Do you plan to have genetic testing?" with response options of yes=1; maybe=2; no=3
Time Frame: Assessed within 1 week after completing the genetic counseling session
Population: The analysis included clients who were offered genetic testing in the session and completed the post-genetic counseling session survey. Two clients, one in each arm, were not offered genetic testing.
Measure: Count of Participants; unit: Participants
Groups:
- Self-affirmation (SA) Group: Immediately prior to the scheduled cancer genetic counseling appointment, clients:
  1. completed standardized questionnaires on self-affirmation (SA) intervention that focused on positive values of personal importance. The SA intervention required clients to rank 11 items (artistic skills, athletics, business/money, creativity, independence, music, politics, relationships with friends and family, religious values, sense of humor, spontaneity) from most important to least important and to elaborate on one that was most important to them and why;
  2. 6-item standardized measure of anxiety questionnaire;
  3. after the counseling session, clients were required to fill out a post session questionnaire
Arm/Group | Self-affirmation (SA) Group | Control Group
Number analyzed (Participants) | 18 | 16
Participants
  Response = Yes | 14 | 15
  Response = No | 2 | 0
  Response = Maybe | 2 | 1

2. Primary Outcome: Number of Clients Who Indicated "Intention to Talk With Family" About Genetic Testing Result
Description: Intention to talk with family was measured with a single categorical survey item, "Which best describes your plans to talk with your family members about genetic testing results (check the one answer that is most true for you)?"
Time Frame: Assessed within 1 week after completing the genetic counseling session
Population: The analysis included clients who completed the post-genetic counseling session survey
Measure: Count of Participants; unit: Participants
Arm/Group | Self-affirmation (SA) Group | Control Group
Number analyzed (Participants) | 19 | 17
Participants
  "I don't plan to talk to anyone" | 0 | 0
  "I plan to talk to only a few people who are closest to me" | 1 | 1
  "I plan to talk to some of my family members" | 3 | 2
  "I plan to talk to most of my first and second degree relatives who are at risk for cancer" | 3 | 6
  "I plan to talk to almost all of my first and second degree relatives who are at risk for cancer" | 2 | 0
  "I plan to talk to almost all of my family members" | 10 | 8

3. Primary Outcome: Likelihood of Talking With Family Members
Description: Likelihood of talking with family members was measured with a single survey item on a 7 point scale, "How likely are you to share results with the relatives you selected?" with 1= Extremely unlikely; 7=Extremely likely
Time Frame: Assessed within 1 week after completing the genetic counseling session
Population: The analysis included clients who completed the post-genetic counseling session survey
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Self-affirmation (SA) Group | Control Group
Number analyzed (Participants) | 19 | 17
units on a scale | 6.74 (0.56) | 6.88 (0.33)

4. Primary Outcome: Decision Self-efficacy: Ability to Confidently Make Decision About Genetic Testing
Description: Decision Self-efficacy was measured with the 12 item Decision Self-efficacy Scale by O'Connor, 1995. Scores ranged from 1-5 with higher average scores indicating higher decision self-efficacy
Time Frame: Assessed within 1 week after completing the genetic counseling session
Population: The analysis included clients who completed the post-genetic counseling session survey
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Self-affirmation (SA) Group | Control Group
Number analyzed (Participants) | 19 | 17
units on a scale | 4.95 (0.09) | 4.85 (0.26)

5. Primary Outcome: Client Knowledge: Hereditary Breast and Ovarian Cancer (HBOC) Knowledge Post Counselling Session
Description: Hereditary Breast and Ovarian Cancer (HBOC) Knowledge was measured with an adapted 7-question scale based on the National Center for Human Genome Research Knowledge (NCHGRK) Scale [Scherr et al. 2015; Kaphingst et al. 2012]. All questions in the scale were presented as True/False. Each question in the scale had a correct answer (coded as 1) and incorrect answer (coded as 0). This adapted HBOC Knowledge Scale score was calculated by summing the total value across the seven questions, with a range of 0 (minimum score, all incorrect) to 7 (maximum score, all correct). Higher score indicates higher knowledge.
Time Frame: Assessed within one week after completing the genetic counseling session
Population: The analysis included clients who completed the post-genetic counseling session survey
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Self-affirmation (SA) Group | Control Group
Number analyzed (Participants) | 19 | 17
units on a scale | 5.78 (0.88) | 6.12 (1.05)

6. Primary Outcome: Patient Empowerment (Client Completed): Ability to Manage Information and Risk Associated With Hereditary Breast and Ovarian Cancer (HBOC) (Decisional Control, Cognitive Control, Behavioral Control, Emotional Regulation, and Hope)
Description: Patient empowerment (client completed) was measured with the 24 item Genetic Counseling Outcomes Scale (GCOS-24; McAllister et al, 2011) using 7-point score ranging from 1=strongly disagree to 7= strongly agree. Higher scores indicate higher empowerment.
Time Frame: Assessed within one week after completing the genetic counseling session
Population: The analysis included clients who completed the post-genetic counseling session survey
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Self-affirmation (SA) Group | Control Group
Number analyzed (Participants) | 19 | 17
units on a scale | 5.86 (0.65) | 5.83 (0.67)

7. Primary Outcome: Patient Empowerment (Genetic Counselor Completed): Client's Ability to Manage Information and Risk Associated With HBOC (Decisional Control, Cognitive Control, Behavioral Control, Emotional Regulation, and Hope)
Description: Patient empowerment (genetic counselor completed) was measured with the 24 item Genetic Counseling Outcomes Scale (GCOS-24; McAllister et al, 2011) using 7-point score ranging from 1=strongly disagree to 7= strongly agree. Higher scores indicate higher empowerment
Time Frame: Assessed immediately after completing the genetic counseling visit
Population: The genetic counselor analysis included all clients who had a genetic counseling session
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Self-affirmation (SA) Group | Control Group
Number analyzed (Participants) | 23 | 22
units on a scale | 5.69 (0.51) | 5.73 (0.59)

8. Secondary Outcome: Mammogram Intention After Counseling: Likelihood of Getting a Mammogram
Description: Mammogram intention was measured with a single survey item on a 7 point scale "How likely are you to get regular mammograms?" with 1= Extremely unlikely to 7=Extremely likely
Time Frame: Assessed within one week after completing the genetic counseling session
Population: The analysis included clients who completed this item on the post-genetic counseling session survey. Two clients, one from each group, skipped the item.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Self-affirmation (SA) Group | Control Group
Number analyzed (Participants) | 18 | 16
units on a scale | 6.78 (1.71) | 6.94 (0.25)

9. Secondary Outcome: Client Anxiety After Writing Exercise and Prior to Counseling
Description: Patient anxiety was measured using the 6 item short version of the Spielberger State Anxiety Scale, a 4-point scale; 1= not at all, 2=somewhat, 3=moderately, 4= very much. Higher score indicates higher anxiety
Time Frame: Assessed immediately after completing the writing exercise and prior to the genetic counseling session
Population: The analysis included clients who completed the writing activity. One client in the control group skipped the item.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Self-affirmation (SA) Group | Control Group
Number analyzed (Participants) | 23 | 21
units on a scale | 2.54 (0.77) | 2.43 (0.81)

10. Secondary Outcome: Perceived Effect of Writing Exercise on Genetic Counseling Visit: Number of Clients With Perceived Effect of Intervention After Writing Exercise
Description: Perceived effect of writing exercise on genetic counseling visit was measured using a single item "The values writing activity affected my appointment"; 1=yes; 2=no
Time Frame: Assessed within one week after completing the genetic counseling session
Population: The analysis included clients who completed the post-genetic counseling session survey
Measure: Count of Participants; unit: Participants
Arm/Group | Self-affirmation (SA) Group | Control Group
Number analyzed (Participants) | 19 | 17
Participants
  Response = Yes | 0 | 0
  Response = No | 19 | 17

11. Secondary Outcome: Perception That Writing Exercise Hindered Genetic Counseling Visit: Number of Clients
Description: Perception that writing exercise hindered the genetic counseling visit was measured using a single survey item "The values writing activity hindered my interaction with my genetic counselor"; 1=yes; 2=no
Time Frame: Assessed within one week after completing the genetic counseling session
Population: The analysis included clients who completed the post-genetic counseling session survey
Measure: Count of Participants; unit: Participants
Arm/Group | Self-affirmation (SA) Group | Control Group
Number analyzed (Participants) | 19 | 17
Participants
  Response = Yes | 0 | 0
  Response = No | 19 | 17

12. Secondary Outcome: Perception That Intervention Improved Genetic Counseling Visit: Number of Clients
Description: Perception that intervention improved the genetic counseling visit was measured using a single survey item "The values writing activity improved my interaction with my genetic counselor"; 1=yes; 2=no
Time Frame: Within 1 week after completing the genetic counseling session
Population: The analysis included clients who completed the post-genetic counseling session survey
Measure: Count of Participants; unit: Participants
Arm/Group | Self-affirmation (SA) Group | Control Group
Number analyzed (Participants) | 19 | 17
Participants
  Response = Yes | 6 | 3
  Response = No | 13 | 14

13. Secondary Outcome: Level of Engagement With the Writing Exercise: Number of Words in Writing Intervention
Description: Number of words in writing intervention was measured by counting the number of words in the essay written by the client
Time Frame: At the time of the intervention
Population: The analysis included clients who completed the writing intervention. Two clients skipped the item.
Measure: Mean (Standard Deviation); unit: words
Arm/Group | Self-affirmation (SA) Group | Control Group
Number analyzed (Participants) | 23 | 20
words | 57.0 (45.7) | 26.2 (15.3)

14. Secondary Outcome: Level of Engagement With the Writing Exercise: Number of Words in Writing Intervention Discussing Importance of Selected Value
Description: Number of Words in Writing Intervention Discussing Importance of Selected Value was measured by counting the number of words in the essay written by the client that were in phrases that were focused on discussing the importance of the selected value, as coded by two coders.
Time Frame: At the time of the intervention
Population: The analysis included clients who completed the writing intervention. Two clients skipped the item.
Measure: Mean (Standard Deviation); unit: words
Arm/Group | Self-affirmation (SA) Group | Control Group
Number analyzed (Participants) | 23 | 20
words | 13.4 (12.1) | 11.4 (10.0)

15. Secondary Outcome: Level of Engagement With the Writing Exercise: Number of Words in Writing Intervention Discussing How Value Was Recently Used
Description: Number of Words in Writing Intervention Discussing How Value Was Recently Used was measured by counting the number of words in the essay written by the client that were in phrases that were focused on discussing how the value was recently used.
Time Frame: At the time of the intervention
Population: The analysis included clients who completed the writing intervention. Two clients skipped the item.
Measure: Mean (Standard Deviation); unit: words
Arm/Group | Self-affirmation (SA) Group | Control Group
Number analyzed (Participants) | 23 | 20
words | 32.5 (33.8) | 3.8 (6.6)

16. Secondary Outcome: Level of Engagement With the Writing Exercise: Number of Examples of How Value Was Recently Used
Description: Number of Examples of How Value was Recently Used was measured by counting the number of unique examples offered in the essay as coded by two coders.
Time Frame: At the time of the intervention
Population: The analysis included clients who completed the writing intervention. Two clients skipped the item.
Measure: Mean (Standard Deviation); unit: unique examples
Arm/Group | Self-affirmation (SA) Group | Control Group
Number analyzed (Participants) | 23 | 20
unique examples | 1.6 (1.4) | 0.2 (0.4)

17. Secondary Outcome: Level of Engagement With the Writing Exercise: Essay Attitude Strength
Description: Essay Attitude Strength is a measure of the extent to which the participant's essay demonstrated the importance of the value selected during the writing exercise. Two independent raters read a subset of the essays and used a scoring system based on the procedure described in Harris & Napper (2005). Each rater gave the participant's essay a numeric score between 1 and 7, and the two scores were examined for inter-rater reliability. The primary rater then rated the remaining essays and the final score was the rating assigned by the primary rater for all essays. A score of 1 (minimum) indicated that the selected value appeared to be not at all important to the participant. A score of 7 (maximum) indicated that the selected value appeared to be very important to the participant.
Time Frame: At the time of the intervention
Population: The analysis included clients who completed the writing intervention. Two clients skipped the item.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Self-affirmation (SA) Group | Control Group
Number analyzed (Participants) | 23 | 20
units on a scale | 5.4 (2.5) | 2.3 (1.3)

18. Secondary Outcome: Level of Engagement With the Writing Exercise: Self-affirmation Score
Description: Self-affirmation score is a measure of the extent to which the essay appeared to be self-affirming for the participant. Two independent raters scored a subset of essays using a system based on procedures described in Harris & Napper (2005) and Ferrer et al. (2017) using the following instructions: "Setting aside your own opinions and values, how self-affirmed would you estimate the writer of this passage to have been (at the end)?" Raters scored each essay and the two scores were examined for inter-rater reliability. The primary rater then rated the remaining essays and the final score was the rating assigned by the primary rater for all essays. A score of 1 (minimum) indicated the value was important but did not include descriptions of why the value was important to the participant. A control group participant received a score of 1 if they followed the writing activity's instructions exactly. A score of 5 (maximum) indicated that the essay elaborated on why the value was important.
Time Frame: At the time of the intervention
Population: The analysis included clients who completed the writing intervention. Two clients skipped the item.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Self-affirmation (SA) Group | Control Group
Number analyzed (Participants) | 23 | 20
units on a scale | 3.7 (1.2) | 1.7 (1.0)

ADVERSE EVENTS:
Time Frame: 1 day
Groups:
- Control Group: Immediately prior to the scheduled cancer genetic counseling appointment, clients:
  1. completed similar standardized questionnaire as the SA group, but was a non-affirming exercise. The non-intervention required clients to rank 11 items (artistic skills, athletics, business/money, creativity, independence, music, politics, relationships with friends and family, religious values, sense of humor, spontaneity) from most important to least important and to elaborate on the 9th ranked item and why it might be important to someone else;
  2. 6-item standardized measure of anxiety questionnaire;
  3. after the counseling session, clients were required to fill out a post session questionnaire
Arm/Group | Self-affirmation (SA) Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/22
Other Adverse Events (participants affected / at risk) | 0/23 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-30): https://cdn.clinicaltrials.gov/large-docs/70/NCT03225170/Prot_SAP_000.pdf